CLINICAL TRIAL: NCT03118895
Title: A Study Evaluating the Safety and Efficacy of the BioFreedom™ Biolimus A9™ Coated Cobalt Chromium Coronary Stent System in Patients at High Risk of Bleeding
Brief Title: Leaders Free III: BioFreedom™ Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosensors Europe SA (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17EU01
Record Dates: First submitted 2017-04-09; First posted 2017-04-18 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Cardiac Death; Myocardial Infarction; Stent Thrombosis; Bleeding; Mortality
MeSH Terms: conditions — Death; Myocardial Infarction; Hemorrhage

STUDY DESIGN:
Masking Description: 370 high bleeding risk items
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Patients with coronary artery disease at high risk of bleeding receiving the BioFreedom™ BA9™ drug-coated stent
  Interventions: Device: BioFreedom™ BA9™ drug-coated stent

INTERVENTIONS:
Device: BioFreedom™ BA9™ drug-coated stent — Drug-coated stent for coronary arteries

SUMMARY:
A study evaluating the safety and efficacy of the BioFreedom™ Biolimus A9™ coated Cobalt Chromium coronary stent system in patients at high risk of bleeding

DETAILED DESCRIPTION:
Prospective, multi-center, open-label single-arm study designed to enroll 370 HBR patients (for at least 340 evaluable) at up to 20 centers in up to 2 European countries. 370 patients will receive a BioFreedomTM CoCr stent. All patients will be followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients at high bleeding risk (HBR) with an indication for percutaneous coronary intervention who can tolerate no more than one month of DAPT. This includes candidates with stable angina, silent ischemia, ACS (STEMI and non-STEMI), non-native lesions and in-stent restenosis. Patients must provide written informed consent.

Reasons of unsuitability for > 1 month dual antiplatelet treatment must include one or MORE of the following:

1. Adjunctive oral anticoagulation treatment planned to continue after PCI
2. Age ≥ 75 years old
3. Baseline Hgb <11 g/dl (or anemia requiring transfusion during the 4 weeks prior to inclusion into the trial)
4. Any prior intracerebral bleed
5. Any stroke in the last 12 months
6. Hospital admission for bleeding during the prior 12 months
7. Non skin cancer diagnosed or treated ≤ 3 years
8. Planned daily NSAID (other than aspirin) or steroids for ≥ 30 days after PCI
9. Planned surgery that would require interruption of DAPT (within next 12 months)
10. Renal failure defined as: Creatinine clearance <40 ml/min
11. Thrombocytopenia (PLT <100,000/mm3)
12. Severe chronic liver disease defined as: patients who have developed any of the following: variceal hemorrhage, ascites, hepatic encephalopathy or jaundice
13. Expected non-compliance to prolonged DAPT for other medical reasons

Exclusion Criteria:

1. Pregnant and breastfeeding women
2. Patients expected not to comply with 1 month DAPT
3. Patients requiring a planned staged PCI procedure more than one week after the index procedure
4. Procedure requires the use of non-study stents, or alternative therapeutic options not followed by stent implantation (angioplasty only, atherectomy only).
5. Active bleeding at the time of inclusion
6. If patient requires a stent <2.5mm
7. If patient requires a stent >3.5mm
8. Cardiogenic shock
9. Compliance with long-term single anti-platelet therapy unlikely
10. Known hypersensitivity or contraindication to aspirin, clopidogrel (or to any another P2Y12 inhibitor if applicable), cobalt chromium, zinc, Biolimus A9TM or a sensitivity to contrast media, which cannot be adequately pre-medicated
11. PCI during the previous 12 months for a lesion other than the target lesion
12. Participation in another clinical trial (12 months after index procedure)
13. Patients with a life expectancy of < 1 year

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 404 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
MACE: composite of cardiac death, myocardial infarction and definite/probable stent thrombosis (safety) | at 1 year
  Incidence
clinically driven target lesion revascularization (efficacy) | at 1 year
  incidence

SECONDARY OUTCOMES:
All-cause mortality | At 1 and 4 months, and 1 and 2 years
  incidence
Clinically Driven Target Lesion Revascularization | At 1 and 4 months, and 2 years
  Incidence
Clinically Driven Target Vessel Revascularization | At 1 and 4 months, and 2 years
  Incidence

CONTACTS AND LOCATIONS:
Overall Officials: Franz Eberli, Prof., Principal Investigator — Chief of Cardiology - Triemli Hospital Zurich - Switzerland; Philippe Garot, MD, Principal Investigator — Hôpital Privé Claude Galien ICPS - France
Locations (2):
- at Hôpital Privé Claude Galien ICPS, Quincy-sous-Sénart, Essonne, France
- Triemli Stadtspital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eberli FR, Oldroyd KG, Urban P, Krucoff MW, Morice MC, Tanguay JF, Leon MB, Brunel P, Maillard L, Lipiecki J, Cook S, Berland J, Hovasse T, Carrie D, Schutte D, Sadozai Slama S, Garot P. Clinical outcomes with thin versus thick strut polymer-free biolimus-coated stents at 3 years. Open Heart. 2024 Jun 18;11(1):e002679. doi: 10.1136/openhrt-2024-002679. PMID 38890129